CLINICAL TRIAL: NCT01026480
Title: Ileal Pouch-Anal Anastomosis (IPAA) Registry
Brief Title: Ileal Pouch-Anal Anastomosis Registry
Acronym: IPAA
Status: Terminated | Type: Observational
Why Stopped: Researchers leading this study have left BMC
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Francis Farraye, MD, Faculty member, Boston Medical Center
Other Study IDs: H-28518
Record Dates: First submitted 2009-11-25; First posted 2009-12-04 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Ileal Pouch-Anal Anastomosis
Keywords: Ileal Pouch Anal Anastomosis; IPAA; Pull through; IBD; Ulcerative colitis; Familial adenomatous polyposis; FAP; Hereditary nonpolyposis colorectal cancer; HNPCC
MeSH Terms: conditions — Colitis, Ulcerative; Adenomatous Polyposis Coli; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IPAA Patients: Patients who have had their IPAA procedures performed by Dr. Becker

SUMMARY:
Little is known about the factors that predispose patients to complications after an ileal pouch-anal anastomosis procedure (IPAA). Our goal is to establish a registry that prospectively captures pre- and post-surgical data from participants. Retrospective studies concerning IPAA outcomes and will be conducted using these data.

DETAILED DESCRIPTION:
In order to better understand the long-term outcomes following IPAA, a registry that collects pertinent information about the underlying disease and its treatments and complications in an organized manner must be established. Establishing this Registry will allow us to follow patients who have an IPAA and organize retrospective medical information into a meaningful system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with one of the following: Ulcerative colitis, Crohn's disease, Indeterminate colitis, Familial adenomatous polyposis, Hereditary nonpolyposis colorectal cancer, Lynch syndrome I or II, or Gardners' syndrome
* Treated by a Center for Digestive Disorders physician
* Scheduled for, or has undergone, ileal pouch-anal anastomosis procedure

Exclusion Criteria:

* Patients who do not speak a language for which the IRB has approved an Informed Consent Form or Short Form
* Patients who are currently incarcerated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for, or who have undergone, ileal pouch-anal anastomosis (IPAA) procedure and have been treated by a Center for Digestive Disorders physician at Boston Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 936 (Actual)
Dates: Start 2009-11; Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Pouch status: functional pouch or non-functional pouch (diverted or excised) | Once per year for duration of the study
  Participants will be queried once per year as to the status of their intestinal pouch. Patients will have either a functional pouch or a non-functional pouch. A pouch will be considered functional if patient is not temporarily or permanently diverted to an ileostomy.

SECONDARY OUTCOMES:
Quality of life | Once per year for duration of the study
  Participants will be queried once per year as to their quality of life using the IBDQ-10.
Health status | Once per year for duration of the study
  Participants will be queried once per year regarding health issues with pouch such as pouchitis, stricture and fistula. Participants will also be asked about presence of co-morbidities such as hypertension, diabetes and arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: James M Becker, MD, Principal Investigator — Boston Medical Center; Francis A Farraye, MD, Study Director — Boston Medical Center; Arthur F Stucchi, PhD, Study Director — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: IPAA Registry at Boston Medical Center — http://www.bmc.org/ipaa/registry.htm